CLINICAL TRIAL: NCT02603042
Title: Biomarker for Hypophosphatasia Disease AN INTERNATIONAL, MULTICENTER, EPIDEMIOLOGICAL PROTOCOL
Brief Title: Biomarker for Hypophosphatasia Disease (BioHypophos)
Acronym: BioHypophos
Status: Withdrawn | Type: Observational
Why Stopped: Transition to BioMetabol
Sponsor: CENTOGENE GmbH Rostock (Industry)
Responsible Party: Sponsor
Other Study IDs: BHP 06-2018
Record Dates: First submitted 2015-11-10; First posted 2015-11-11 (Estimated); Last update posted 2023-02-13 (Actual); Status verified 2023-02

CONDITIONS: Defective Mineralization
Keywords: Hypophosphatasia Disease; Biomarker

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — For the development of the new biomarkers using the technique of Mass-spectrometry 7, 5 ml EDTA blood and a dry blood spot filter card are taken. To proof the correct di- agnosis of Hypophosphatasia in those patients where up to the enrollment in the study no genetic testing has been done, sequencing of Hypophosphatasia disease will be done. The analyses will be done at the: Centogene AG Am Strande 7 18055 Rostock Germany
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Observation: Patients with Hypophosphatasia disease or high-grade suspicion for Hypophosphatasia disease

SUMMARY:
Development of a new MS-based biomarker for the early and sensitive diagnosis of Hypophosphatasia disease from plasma

DETAILED DESCRIPTION:
Hypophosphatasia (HPP) is a rare genetic disorder characterized the abnormal development of bones and teeth. These abnormalities occur due to defective mineralization, the process by which bones and teeth take up minerals such as calcium and phosphorus. These minerals are required for proper hardness and strength. Defective mineralization results in bones that are soft and prone to fracture and deformity. Defective mineralization of teeth can lead to premature tooth loss. The specific symptoms can vary greatly from one person to another, sometimes even among members of the same family. There are five major clinical forms of HPP that range from an extremely severe form that can cause stillbirth to a form associated with only premature loss of baby (deciduous) teeth, but no bone abnormalities. Hypophosphatasia is caused by mutations in the tissue non-specific alkaline phosphatase (ALPL) gene. This gene is also known as the TNSALP gene. Such mutations lead to low levels of the tissue nonspecific alkaline phosphatase enzyme. Depending on the specific form, hypophosphatasia can be inherited in an autosomal recessive or autosomal dominant manner.

Hypophosphatasia is an extremely variable disorder. Five major clinical forms have been identified based primarily upon the age of onset of symptoms and diagnosis. These are known as perinatal, infantile, childhood, adult, and odontohypophosphatasia. Generally, the severity of these different forms of hypophosphatasia correlates to the residual alkaline phosphate activity in the body, with less enzyme activity causing more severe dis- ease. Because hypophosphatasia is a highly variable disorder, it is important to note that affected individuals may not have all of the symptoms and that every individual case is unique. Some children will develop severe complications early in life; others have mild disease that may improve during young adult life.

Perinatal hypophosphatasia is associated with profound inactivity of alkaline phosphatase and markedly impaired mineralization. Consequently, the skeleton fails to form properly in the womb. Specific skeletal malformations may vary, but short, bowed arms and legs and underdeveloped ribs often occur. Some pregnancies end in stillbirth. In other cases, affected newborns survive for several days, but pass away from respiratory failure due to deformities of the chest and underdeveloped lungs.

Infantile hypophosphatasia may have no noticeable abnormalities at birth, but symptoms may become apparent at any time within the first six months. The initial symptom may be the failure to gain weight and grow at the expected rate for age and gender referred to as "failure to thrive." Some affected babies later exhibit early fusion of the bones of the skull (craniosynostosis), which can result in the head appearing disproportionately wide (brachycephaly). Craniosynostosis may be associated with increased pressure of the cerebrospinal fluid, a condition known as "intracranial hypertension." This complication can cause headaches, swelling of the optic disk (papilledema), and bulging of the eyes (proptosis). Affected infants have softened, weakened bones that lead to the skeletal malformations of rickets. Rickets is a bone disease that occurs during growth with softening of bone and characteristic bowing deformities of the legs from growth plate abnormalities. Enlarged wrist and ankle joints may occur. Affected infants may also have deformities in the chest and ribs and rib fractures, predisposing them to pneumonia. Varying degrees of pulmonary insufficiency and breathing difficulties may develop, potentially progressing to life-threatening respiratory failure. Episodes of fever and bone pain, or tender bones may occur. Some infants exhibit diminished muscle tone (hypotonia) so that a baby appears "floppy" as well as elevated levels of calcium in the blood (hypercalcemia). Hypercalcemia can cause vomiting, constipation, weakness, and poor feeding. In rare cases, vitamin B6-dependent seizures may occur. Increased excretion of calcium may lead to kidney (renal) damage. Sometimes there is spontaneous improvement in mineralization during early childhood, with the exception of craniosynostosis. Short stature and skeletal deformities may persist lifelong.

Childhood hypophosphatasia is highly variable, but is less severe than the infantile form. Affected children may sometimes have craniosynostosis and exhibit signs of intra- cranial hypertension. Skeletal malformations that resemble rickets may become apparent at 2 to 3 years of age. Bone and joint pain and fractures may occur. Baby teeth may fall out earlier than normal. Some children are weak and experience delays in walking, and when they do learn to walk may have a distinct, waddling gait. Spontaneous remission of bone symptoms has been reported in young adult life, but such symptoms can recur during middle age or late adulthood.

Adult hypophosphatasia is characterized by a wide variety of symptoms. Affected individuals have osteomalacia, a softening of the bones in adults. Some individuals have a history of rickets during childhood, or have experienced premature loss of their baby teeth. Individuals with adult hypophosphatasia can experience fractures, especially stress fractures in the feet or pseudofractures of the thigh. Repeated fractures can result in chronic pain and debility. Fractures of the spine seem less common, but also occur. Bone pain is a common complication. Some affected adults develop joint inflammation and pain near or around certain joints due to the accumulation of calcium crystals (calcific periarthritis) or a condition called chondrocalcinosis, characterized by the accumulation of calcium crystals within the cartilage of joints, sometimes damaging the joint. Others have sudden, severe pain in the joint (pseudo gout). Affected adults may experience loss of adult teeth.

Odontohypophosphatasia is characterized by the premature loss of teeth in childhood, or loss of teeth in adulthood. It is an isolated finding that does not occur along with the characteristic bone symptoms of other forms of hypophosphatasia.

For hypophosphatasia, mutations in the ALPL gene can be inherited in an autosomal recessive or autosomal dominant manner. The perinatal and infantile forms of HPP are inherited in an autosomal recessive manner. The childhood form can be autosomal recessive or autosomal dominant. The adult form and odontohypophosphatasia typically are autosomal dominant disorders, but in rare cases can be inherited as an autosomal recessive trait.

A diagnosis of hypophosphatasia is based upon identification of characteristic signs and symptoms, a detailed patient history, a thorough clinical evaluation, and a variety of laboratory tests including x-ray studies. Proper diagnosis of hypophosphatasia is easy for physicians who are familiar or experienced with this disorder.

New methods, like mass-spectrometry give a good chance to characterize specific metabolic alterations in the blood (plasma) of affected patients that allow diagnosing in the future the disease earlier, with a higher sensitivity and specificity.

Therefore it is the goal of the study to identify and validate a new biochemical marker from the plasma of the affected patients helping to benefit other patients by an early diagnose and thereby with an earlier treatment.

ELIGIBILITY:
IInclusion Criteria:

* Informed consent will be obtained from the patient or the parents before any study related procedures.
* Patients of both genders older than 2 month
* The patient has a diagnosis of Hypophosphatasia disease or a high-grade suspicion for Hypophosphatasia disease
* High-grade suspicion present, if one or more inclusion criteria are valid:

  * Positive family anamnesis for Hypophosphatasia disease
  * Frequent fractures
  * Bone pain
  * Tooth loss
  * Osteopenia/Osteoporosis
  * Craniosynostosis

Exclusion Criteria:

* No Informed consent from the patient or the parents before any study related procedures.
* Patients of both gender younger than 2 month
* No diagnosis of Hypophosphatasia disease or no valid criteria for profound suspicion of Hypophosphatasia disease

Min Age: 2 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with Hypophosphatasia disease or high-grade suspicion for Hypophosphatasia disease
Sampling Method: Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2018-08-20 (Actual); Primary Completion 2021-02-28 (Actual); Study Completion 2021-02-28 (Actual)

PRIMARY OUTCOMES:
Sequencing of the Hypophosphatasia disease related gene | 4 weeks
  Next-Generation Sequencing (NGS) of the ALPL gene will be performed. The mutation will be confirmed by Sanger sequencing.

SECONDARY OUTCOMES:
The Hypophosphatasia disease specific biomarker candidates finding | 24 months
  The quantitative determination of small molecules (molecular weight 150-700 kD, given as ng/μl) within a dried blood spot sample will be validated via liquid chromatography multiple reaction-monitoring mass spectrometry (LC/MRM-MS) and compared with a merged control cohort. The statistically best validated molecule will be considered as a disease specific biomarker.

CONTACTS AND LOCATIONS:
Locations (3):
- Centogene AG, Rostock, Germany
- NIRMAN Navi Mumbai Institute of Research In Mental And Neurological Handicap/Pediatric Geneticist, Mumbai, India
- Lady Ridgeway Hospital for Children, Colombo, Sri Lanka

IPD SHARING:
Plan to Share IPD: Undecided